CLINICAL TRIAL: NCT02969356
Title: An International, Multicentre, Prospective, Single-Arm Study to Assess the Effect on Voluntary Movements of AbobotulinumtoxinA 1500 U Administered in Both Upper and Lower Limbs in Conjunction With a Guided Self-Rehabilitation Contract in Adult Subjects With Spastic Hemiparesis
Brief Title: Study to Evaluate Effects of DYSPORT® Injected in Lower and Upper Limb Combined With Guided Self-Rehabilitation Contract (GSC)
Acronym: ENGAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-FR-52120-228; 2016-001989-29 (EudraCT Number)
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Spastic Hemiparesis
MeSH Terms: conditions — Hemiplegia | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dysport (Experimental): Each subject will undergo two intramuscular injection (treatment) cycles, receiving AbobotulinumtoxinA (Dysport®) 1500 U on Day 1 of each cycle; the two dosing occasions will be separated by at least 12 weeks (maximum 20 weeks). Subjects will also receive daily GSC therapy. The main focus of GSC will be on the primary treatment target (TT) limb (as determined at the Baseline Visit) and then the other limb. All muscle groups requiring active training and/or stretching should be trained. Subjects will be be given a diary to record each day whether they have performed the GSC therapy.
  Interventions: Biological: Botulinum toxin type A; Other: GSC

INTERVENTIONS:
Biological: Botulinum toxin type A — Dysport® administered in both upper and lower limbs (total dose of 1500 U per injection split between the 2 limbs).
  Other Names: AbobotulinumtoxinA (Dysport®)
Other: GSC — The GSC is a motivational tool. The physiotherapist will teach each subject the stretching postures and exercises to perform on a daily basis throughout the study. These will be tailored to the individual subject's needs and will form the GSC therapy.

SUMMARY:
The purpose of this clinical study is to assess whether AbobotulinumtoxinA (Dysport®) injections in upper and lower limbs accompanied with a personal exercise plan called "Guided Self-rehabilitation Contract" (GSC) can improve voluntary movements in subjects with hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged at least the national legal adult age.
* Subjects with hemiparesis due to acquired brain injury (ABI) presenting with muscle overactivity impeding motor function based on investigator's judgement including, but not limited to, at least one of the following requiring botulinum neurotoxin (BoNT) treatment: typical clenched fist; flexed wrist; flexed elbow; or plantar flexed foot pattern.
* At least 12 months since the ABI (i.e. stroke or traumatic brain injury (TBI)).
* Naïve or non-naïve to BoNT treatment; if non-naïve, at least 4 months after the last BoNT injection, of any serotype.
* Upper limb active function with an overall score between 2 and 7, as assessed by Modified Frenchay Scale (MFS), if the primary TT limb is the upper limb (UL).
* A 10-metre maximal WS barefoot between 0.2 and 1.4 m/s, if the primary TT limb is the lower limb (LL). Maximal WS barefoot will be performed without walking aids. However, a cane may be permitted if absolutely necessary (although this may prevent detection of treatment-induced improvements). In this case, the same aid will have to be used for all WS assessments during the study.
* Subjects must provide written informed consent to participate in the study prior to any study-related procedures.
* Female subjects of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study until the last visit of the subjects and for at least 12 weeks post injection. Acceptable methods of contraception include total abstinence, male partner has had a vasectomy, double barrier method (e.g. male condom plus spermicide, or female diaphragm plus spermicide), intrauterine device, or hormonal contraceptive (oral, transdermal, implanted and injected).
* Subjects must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period and willing to return to the clinic for the follow-up evaluation as specified in the protocol

Exclusion Criteria:

* Inability to understand protocol procedures and requirements, which, in the opinion of the investigator, could negatively impact on protocol compliance, in particularly inability to exercise according to the GSC.
* Previous surgery on the affected muscles and ligaments, tendons, nerve trunks, or bones of the treated upper or lower limb.
* Previous treatment with phenol and/or alcohol in any of the treated limbs any time before the study.
* Any medical condition (including severe dysphagia or breathing difficulties) that may increase, in the opinion of the investigator, the likelihood of adverse events (AEs) related to BoNT A treatment.
* Current, planned or received within the last 4 weeks prior to study treatment, treatment with any drug that interferes either directly or indirectly with neuromuscular function (for example, aminoglycosides).
* Major neurological impairment other than spastic paresis (including major proprioceptive ataxia or apraxia on the paretic side) that could negatively impact on the functional performance of the subject.
* Known disease of the neuromuscular junction (such as Lambert-Eaton myasthenic syndrome or myasthenia gravis).
* Known sensitivity to BoNT-A or any excipient of Dysport.
* Infection at the injection site(s).
* Current pregnancy or lactation. A pregnancy test will be performed at the start of the study for all female subjects of childbearing potential (i.e. not surgically sterile or 2 years postmenopausal).
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude.
* Abnormal baseline findings or any other medical condition(s) that, in the opinion of the investigator, might jeopardise the subject's safety.
* Subjects treated, or likely to be treated, with intrathecal baclofen during the course of the study or during the 4 weeks before study entry.
* Subjects who have participated in any therapeutic clinical study/received any investigational agent within 30 days of enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-12-18; Primary Completion 2018-04-26 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (19):
- United States (6):
  - Kansas Institute of Research, Kansas City Bone & Joint Clinic, Division of Signature Medical Group of KC, Kansas City, Kansas
  - University of Pittsburgh Medical Center, Physical Medicine and Rehabilitation, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Department of Neurology, Division of Movement Disorders, Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Health Physical Medicine & Rehabilitation Department, TIRR Memorial Hermann, Houston, Texas
- Czechia (5):
  - Fakultní nemocnice Královské Vinohrady, Neurologická klinika, Brno
  - Neurology and Physiotherapy Outpatient Clinic, Brno
  - Fakultní nemocnice Brno Neurologická klinika, Brno
  - Neurology Department - Regional Hospital Pardubice, Pardubice
  - Department of Neurology and Center of Clinical Neuroscience, Charles University in Prague, 1st Faculty of Medicine and General University Hospital in Prague, Prague
- France (4):
  - Service de Médecine Physique et Réadaptation, Hôpital Albert-Chenevier, Créteil, Cedex
  - Service de Médecine Physique et de Réadaptation, Bâtiment Tastet-Girard, Groupe Hospitalier Pellegrin, Bordeaux
  - Service de Médecine Physique et Réadaptation, Hôpital Sébastopol - CHU de Reims, Reims
  - Service de Médecine Physique et Réadaptation, CHU Saint Etienne - Hôpital Bellevue, Saint-Etienne
- Russia (4):
  - Federal Siberian Scientific Clinical Center, Krasnoyarsk
  - Medical Rehabilitation Center, Moscow
  - Saint-Petersburg Bekhterev Psychoneurological Research Institute, Saint Petersburg
  - Samara Regional Clinical Hospital n.a. V.D.Seredavin, Samara

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Gracies JM, Francisco GE, Jech R, Khatkova S, Rios CD, Maisonobe P; ENGAGE Study Group. Guided Self-rehabilitation Contracts Combined With AbobotulinumtoxinA in Adults With Spastic Paresis. J Neurol Phys Ther. 2021 Jul 1;45(3):203-213. doi: 10.1097/NPT.0000000000000359. PMID 34039905
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2023/05/11173817/ENGAGE-Lay-Summary-2020.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, single-arm study was conducted in 18 centers in 4 countries between 22 December 2016 and 18 July 2018 in participants with spastic hemiparesis due to acquired brain injury. Study had 2 treatment cycles separated by at least 12 (maximum 20) weeks and combined with Guided Self-Rehabilitation Contract (GSC) for whole study duration.
Pre-assignment Details: A total of 157 participants were treated in this study. At baseline (Cycle 1, Day 1), the primary treatment target (TT) limb (upper limb [UL] or lower limb [LL]) was defined by the investigator, following discussion with the participant. If the primary TT limb was the UL, the secondary TT limb was the LL (and vice versa).
Groups:
- Dysport: Dysport (AbobotulinumtoxinA) 1500 units (U) intramuscular (IM) injection, was administered as a split dose, in both the UL and LL on Day 1 of each treatment cycle. The dose given in each limb was based on which was considered the primary TT limb at baseline. At least half the total dose must have been injected in the primary TT limb and a maximum of 1000 U could be injected in an UL (even if it was the primary TT limb). There was no maximum dose that could have been injected in a LL, provided that some out of the 1500 U total was used for the UL injection.
  The second Dysport injection (Cycle 2) may have been given in a different split to the first injection (Cycle 1), at the discretion of the investigator. However, the same minimal/maximal rules applied. The primary TT remained the same for both Dysport injections.
  Participants were also asked to perform daily GSC therapy throughout the study.
Period: Overall Study
Arm/Group | Dysport
Started | 157
Intent-to-Treat (ITT) Population | 153
Completed | 134
Not Completed | 23
Not completed — Adverse Event | 7
Not completed — Consent withdrawn | 2
Not completed — Lost to Follow-up | 3
Not completed — Did not need to be reinjected | 6
Not completed — Personal reasons | 5

BASELINE CHARACTERISTICS:
Population: The ITT population included all participants who were injected at least once with the study treatment, who received at least one day of GSC therapy during the study and for whom a primary TT limb had been defined.
Groups:
- Dysport: Dysport 1500 U IM injection, was administered as a split dose, in both the UL and LL on Day 1 of each treatment cycle. The dose given in each limb was based on which was considered the primary TT limb at baseline. At least half the total dose must have been injected in the primary TT limb and a maximum of 1000 U could be injected in an UL (even if it was the primary TT limb). There was no maximum dose that could have been injected in a LL, provided that some out of the 1500 U total was used for the UL injection.
  The second Dysport injection (Cycle 2) may have been given in a different split to the first injection (Cycle 1), at the discretion of the investigator. However, the same minimal/maximal rules applied. The primary TT remained the same for both Dysport injections.
  Participants were also asked to perform daily GSC therapy throughout the study.
Arm/Group | Dysport
Number analyzed (Participants) | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 122
  >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 126
  Race: Black or African American | 7
  Race: Asian | 2
  Race: Missing | 18
  Ethnicity: Not Hispanic/Latino | 135
  Ethnicity: Missing | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responder Participants at Week 6 After the Second Injection, According to Composite Active Range of Motion (AROM) in the Primary TT Limb
Description: Percentage of responder participants according to AROM was measured by goniometer in the primary TT limb, using zero as the theoretical position of minimal stretch for the muscle assessed. Participants were asked to perform the active movement as far as possible against that muscle and the angle was measured. A participant was considered a responder if he/she achieved at least the predefined improvement threshold - larger or equal to 35 degrees in UL or 5 degrees in LL - in the primary TT limb (based on the composite AROM individual change from baseline to Week 6 after the second injection).
Time Frame: At Week 6, Cycle 2
Population: The modified ITT (mITT) population included all participants who were injected at least once with the study treatment, who received at least 1 day of GSC therapy during the study, for whom a primary TT limb had been defined and who had the primary efficacy outcome assessed at Week 6, Cycle 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dysport
Number analyzed (Participants) | 136
percentage of participants | 72.1 [64.0 to 78.9]

2. Secondary Outcome: Percentage of Responder Participants at Week 6 After the First Injection, According to Composite AROM in the Primary TT Limb
Description: Percentage of responder participants according to composite AROM was measured by goniometer in the primary TT limb, using zero as the theoretical position of minimal stretch for the muscle assessed. Participants were asked to perform the active movement as far as possible against that muscle and the angle was measured. A participant was considered a responder if he/she achieved at least the predefined improvement threshold - larger or equal to 35 degrees in UL or 5 degrees in LL - in the primary TT limb (based on the composite AROM individual change from baseline to Week 6 after the first injection).
Time Frame: At Week 6, Cycle 1
Population: The ITT population included all participants who were injected at least once with the study treatment, who received at least 1 day of GSC therapy during the study and for whom a primary TT limb had been defined.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dysport
Number analyzed (Participants) | 153
percentage of participants | 58.2 [50.2 to 65.7]

3. Secondary Outcome: Mean Change From Baseline in AROM Against 10 Prespecified Muscle Groups at Week 6 and Week 12 of Each Treatment Cycle, Reinjection Cycle Visit and Last Study Visit
Description: The AROM was measured by goniometer in the primary TT limb, using zero as the theoretical position of minimal stretch for the muscle assessed. Participants were asked to perform the active movement as far as possible against that muscle and the angle was measured. The angle of joint movement was measured in 10 prespecified muscle groups (injected or noninjected); UL: shoulder extensors (SE), elbow flexors (EF), wrist flexors (WF), extrinsic finger flexors (FF) and pronator teres (PT), LL: soleus (Sol), gastrocnemius (GN), gluteus maximus (GM), hamstrings (HS) and rectus femoris (RF). The reinjection cycle visit corresponds to Week 12, 16 or 20 of injection Cycle 1. The last study visit corresponds to the last post-baseline visit performed by the participant (including the early withdrawal visit).
Time Frame: Week 6 and Week 12 of each treatment cycle, reinjection cycle visit and last study visit
Population: The ITT population included all participants who were injected at least once with the study treatment, who received at least 1 day of GSC therapy during the study and for whom a primary TT limb had been defined. Only participants with data available at each time point are presented.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Dysport
Number analyzed (Participants) | 153
degrees
  UL SE: Week 6, Cycle 1: number analyzed (Participants) | 149
  UL SE: Week 6, Cycle 1 | 8.9 (16.4)
  UL SE: Week 12, Cycle 1: number analyzed (Participants) | 146
  UL SE: Week 12, Cycle 1 | 15.8 (22.9)
  UL SE: Reinjection cycle visit: number analyzed (Participants) | 140
  UL SE: Reinjection cycle visit | 13.4 (22.5)
  UL SE: Week 6, Cycle 2: number analyzed (Participants) | 136
  UL SE: Week 6, Cycle 2 | 19.3 (25.1)
  UL SE: Week 12, Cycle 2: number analyzed (Participants) | 129
  UL SE: Week 12, Cycle 2 | 21.1 (27.7)
  UL SE: Last study visit: number analyzed (Participants) | 152
  UL SE: Last study visit | 19.0 (24.9)
  UL EF: Week 6, Cycle 1: number analyzed (Participants) | 149
  UL EF: Week 6, Cycle 1 | 8.7 (25.5)
  UL EF: Week 12, Cycle 1: number analyzed (Participants) | 146
  UL EF: Week 12, Cycle 1 | 12.0 (27.3)
  UL EF: Reinjection cycle visit: number analyzed (Participants) | 140
  UL EF: Reinjection cycle visit | 10.9 (28.3)
  UL EF: Week 6, Cycle 2: number analyzed (Participants) | 137
  UL EF: Week 6, Cycle 2 | 14.9 (26.2)
  UL EF: Week 12, Cycle 2: number analyzed (Participants) | 130
  UL EF: Week 12, Cycle 2 | 15.4 (28.1)
  UL EF: Last study visit | 13.0 (28.2)
  UL WF: Week 6, Cycle 1: number analyzed (Participants) | 148
  UL WF: Week 6, Cycle 1 | 11.0 (16.3)
  UL WF: Week 12, Cycle 1: number analyzed (Participants) | 144
  UL WF: Week 12, Cycle 1 | 10.9 (20.1)
  UL WF: Reinjection cycle visit: number analyzed (Participants) | 138
  UL WF: Reinjection cycle visit | 9.6 (20.4)
  UL WF: Week 6, Cycle 2: number analyzed (Participants) | 135
  UL WF: Week 6, Cycle 2 | 15.6 (24.3)
  UL WF: Week 12, Cycle 2: number analyzed (Participants) | 129
  UL WF: Week 12, Cycle 2 | 13.6 (22.4)
  UL WF: Last study visit: number analyzed (Participants) | 151
  UL WF: Last study visit | 12.4 (22.3)
  UL FF: Week 6, Cycle 1: number analyzed (Participants) | 148
  UL FF: Week 6, Cycle 1 | 24.1 (37.1)
  UL FF: Week 12, Cycle 1: number analyzed (Participants) | 144
  UL FF: Week 12, Cycle 1 | 20.7 (36.0)
  UL FF: Reinjection cycle visit: number analyzed (Participants) | 138
  UL FF: Reinjection cycle visit | 14.5 (36.7)
  UL FF: Week 6, Cycle 2: number analyzed (Participants) | 136
  UL FF: Week 6, Cycle 2 | 29.5 (43.7)
  UL FF: Week 12, Cycle 2: number analyzed (Participants) | 129
  UL FF: Week 12, Cycle 2 | 27.9 (49.1)
  UL FF: Last study visit: number analyzed (Participants) | 151
  UL FF: Last study visit | 24.5 (44.9)
  UL PT: Week 6, Cycle 1: number analyzed (Participants) | 149
  UL PT: Week 6, Cycle 1 | 9.0 (32.6)
  UL PT: Week 12, Cycle 1: number analyzed (Participants) | 146
  UL PT: Week 12, Cycle 1 | 8.0 (38.0)
  UL PT: Reinjection cycle visit: number analyzed (Participants) | 140
  UL PT: Reinjection cycle visit | 7.4 (37.9)
  UL PT: Week 6, Cycle 2: number analyzed (Participants) | 137
  UL PT: Week 6, Cycle 2 | 11.0 (38.6)
  UL PT: Week 12, Cycle 2: number analyzed (Participants) | 129
  UL PT: Week 12, Cycle 2 | 9.4 (38.4)
  UL PT: Last study visit: number analyzed (Participants) | 152
  UL PT: Last study visit | 8.7 (41.0)
  LL Sol: Week 6, Cycle 1: number analyzed (Participants) | 149
  LL Sol: Week 6, Cycle 1 | 4.7 (9.6)
  LL Sol: Week 12, Cycle 1: number analyzed (Participants) | 145
  LL Sol: Week 12, Cycle 1 | 5.2 (13.8)
  LL Sol: Reinjection cycle visit: number analyzed (Participants) | 139
  LL Sol: Reinjection cycle visit | 4.5 (15.4)
  LL Sol: Week 6, Cycle 2: number analyzed (Participants) | 137
  LL Sol: Week 6, Cycle 2 | 9.3 (17.9)
  LL Sol: Week 12, Cycle 2: number analyzed (Participants) | 130
  LL Sol: Week 12, Cycle 2 | 9.0 (17.0)
  LL Sol: Last study visit: number analyzed (Participants) | 152
  LL Sol: Last study visit | 8.2 (16.4)
  LL GN: Week 6, Cycle 1: number analyzed (Participants) | 149
  LL GN: Week 6, Cycle 1 | 9.0 (14.8)
  LL GN: Week 12, Cycle 1: number analyzed (Participants) | 145
  LL GN: Week 12, Cycle 1 | 9.9 (14.6)
  LL GN: Reinjection cycle visit: number analyzed (Participants) | 139
  LL GN: Reinjection cycle visit | 7.5 (15.0)
  LL GN: Week 6, Cycle 2: number analyzed (Participants) | 137
  LL GN: Week 6, Cycle 2 | 12.6 (16.8)
  LL GN: Week 12, Cycle 2: number analyzed (Participants) | 130
  LL GN: Week 12, Cycle 2 | 11.8 (17.1)
  LL GN: Last study visit: number analyzed (Participants) | 152
  LL GN: Last study visit | 11.9 (17.4)
  LL GM: Week 6, Cycle 1: number analyzed (Participants) | 149
  LL GM: Week 6, Cycle 1 | 5.1 (15.9)
  LL GM: Week 12, Cycle 1: number analyzed (Participants) | 146
  LL GM: Week 12, Cycle 1 | 5.2 (15.2)
  LL GM: Reinjection cycle visit: number analyzed (Participants) | 140
  LL GM: Reinjection cycle visit | 5.1 (14.7)
  LL GM: Week 6, Cycle 2: number analyzed (Participants) | 137
  LL GM: Week 6, Cycle 2 | 6.1 (15.9)
  LL GM: Week 12, Cycle 2: number analyzed (Participants) | 130
  LL GM: Week 12, Cycle 2 | 7.3 (15.2)
  LL GM: Last study visit | 6.6 (16.5)
  LL HS: Week 6, Cycle 1: number analyzed (Participants) | 149
  LL HS: Week 6, Cycle 1 | 0.9 (34.2)
  LL HS: Week 12, Cycle 1: number analyzed (Participants) | 146
  LL HS: Week 12, Cycle 1 | 4.0 (34.7)
  LL HS: Reinjection cycle visit: number analyzed (Participants) | 140
  LL HS: Reinjection cycle visit | 5.6 (30.7)
  LL HS: Week 6, Cycle 2: number analyzed (Participants) | 137
  LL HS: Week 6, Cycle 2 | 8.2 (25.1)
  LL HS: Week 12, Cycle 2: number analyzed (Participants) | 130
  LL HS: Week 12, Cycle 2 | 10.3 (26.3)
  LL HS: Last study visit | 6.8 (31.1)
  LL RF: Week 6, Cycle 1: number analyzed (Participants) | 148
  LL RF: Week 6, Cycle 1 | 4.5 (15.0)
  LL RF: Week 12, Cycle 1: number analyzed (Participants) | 146
  LL RF: Week 12, Cycle 1 | 4.4 (23.1)
  LL RF: Reinjection cycle visit: number analyzed (Participants) | 140
  LL RF: Reinjection cycle visit | 5.1 (25.3)
  LL RF: Week 6, Cycle 2: number analyzed (Participants) | 137
  LL RF: Week 6, Cycle 2 | 8.9 (24.7)
  LL RF: Week 12, Cycle 2: number analyzed (Participants) | 130
  LL RF: Week 12, Cycle 2 | 9.6 (23.4)
  LL RF: Last study visit | 8.6 (23.0)

4. Secondary Outcome: Mean Change From Baseline in Composite AROM Against Injected Muscle Groups (Any of the 10 Prespecified Muscles) at Week 6 and Week 12 of Each Treatment Cycle, Reinjection Cycle Visit and Last Study Visit
Description: Composite AROM (XA) was measured by goniometer in the primary TT limb (either UL or LL, depending on which one has been selected as the primary TT limb), composite AROM in the UL injected muscle groups was calculated as the sum of the AROM in the EF, WF and FF. Composite AROM in the LL injected muscle groups was calculated as the sum of the AROM in Sol and GN.
Time Frame: Week 6 and Week 12 of each treatment cycle, reinjection cycle visit and last study visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Dysport
Number analyzed (Participants) | 153
degrees
  UL: Week 6, Cycle 1: number analyzed (Participants) | 148
  UL: Week 6, Cycle 1 | 43.1 (49.9)
  UL: Week 12, Cycle 1: number analyzed (Participants) | 144
  UL: Week 12, Cycle 1 | 42.8 (56.7)
  UL: Reinjection cycle visit: number analyzed (Participants) | 138
  UL: Reinjection cycle visit | 34.1 (52.8)
  UL: Week 6, Cycle 2: number analyzed (Participants) | 135
  UL: Week 6, Cycle 2 | 59.5 (64.4)
  UL: Week 12, Cycle 2: number analyzed (Participants) | 129
  UL: Week 12, Cycle 2 | 56.3 (66.7)
  UL: Last study visit: number analyzed (Participants) | 151
  UL: Last study visit | 49.3 (63.4)
  LL: Week 6, Cycle 1: number analyzed (Participants) | 149
  LL: Week 6, Cycle 1 | 13.7 (18.3)
  LL: Week 12, Cycle 1: number analyzed (Participants) | 145
  LL: Week 12, Cycle 1 | 15.1 (23.4)
  LL: Reinjection cycle visit: number analyzed (Participants) | 139
  LL: Reinjection cycle visit | 12.0 (24.5)
  LL: Week 6, Cycle 2: number analyzed (Participants) | 137
  LL: Week 6, Cycle 2 | 21.9 (28.8)
  LL: Week 12, Cycle 2: number analyzed (Participants) | 130
  LL: Week 12, Cycle 2 | 20.8 (28.8)
  LL: Last study visit: number analyzed (Participants) | 152
  LL: Last study visit | 20.1 (27.6)

5. Secondary Outcome: Mean Change From Baseline in Full Composite AROM Against 5 UL or 5 LL Muscle Groups, Regardless of Whether the Muscle Groups Were Injected or Not at Week 6 and Week 12 of Each Treatment Cycle, Reinjection Cycle Visit and Last Study Visit
Description: Full composite AROM, regardless of whether the muscle groups was injected or not was measured by goniometer in the primary TT limb. Full Composite AROM in the UL was calculated as the sum of the AROM in the 5 UL muscle groups (SE+EF+WF+FF+PT). Full Composite AROM in the LL was calculated as the sum of the AROM in the 5 LL muscle groups (Sol+GN+GM+HS+RF).
Time Frame: Week 6 and Week 12 of each treatment cycle, reinjection cycle visit and last study visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Dysport
Number analyzed (Participants) | 153
degrees
  UL: Week 6, Cycle 1: number analyzed (Participants) | 148
  UL: Week 6, Cycle 1 | 60.6 (68.4)
  UL: Week 12, Cycle 1: number analyzed (Participants) | 144
  UL: Week 12, Cycle 1 | 66.3 (75.7)
  UL: Reinjection cycle visit: number analyzed (Participants) | 138
  UL: Reinjection cycle visit | 53.9 (69.9)
  UL: Week 6, Cycle 2: number analyzed (Participants) | 134
  UL: Week 6, Cycle 2 | 90.5 (90.1)
  UL: Week 12, Cycle 2: number analyzed (Participants) | 128
  UL: Week 12, Cycle 2 | 87.6 (94.8)
  UL: Last study visit: number analyzed (Participants) | 150
  UL: Last study visit | 77.8 (89.6)
  LL: Week 6, Cycle 1: number analyzed (Participants) | 148
  LL: Week 6, Cycle 1 | 24.4 (42.7)
  LL: Week 12, Cycle 1: number analyzed (Participants) | 145
  LL: Week 12, Cycle 1 | 28.7 (55.9)
  LL: Reinjection cycle visit: number analyzed (Participants) | 139
  LL: Reinjection cycle visit | 28.0 (56.2)
  LL: Week 6, Cycle 2: number analyzed (Participants) | 137
  LL: Week 6, Cycle 2 | 45.1 (58.2)
  LL: Week 12, Cycle 2: number analyzed (Participants) | 130
  LL: Week 12, Cycle 2 | 48.1 (60.4)
  LL: Last study visit: number analyzed (Participants) | 152
  LL: Last study visit | 42.2 (61.7)

6. Secondary Outcome: Mean Change From Baseline in Modified Frenchay Scale (MFS) Overall Score Evaluated Locally and Centrally at Week 12 of Each Treatment Cycle and Last Study Visit
Description: The MFS was used to measure active function in the UL. The MFS consists of 10 tasks, each of which was evaluated locally by the site investigator and centrally by a blinded central reviewer at the coordinating investigators' site, on a 10-point visual analogue scale (VAS) ranging from "No movement" to "Normal". Higher score indicates a better outcome. The MFS overall scores were obtained by averaging all individual task scores, provided that at least 8 out of the 10 were not missing. The mean change from baseline was calculated for the local and central assessments and a positive change from baseline indicates an improvement in active function.
Time Frame: Week 12 of each treatment cycle and last study visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 153
units on a scale
  Local assessment: Week 12, Cycle 1: number analyzed (Participants) | 141
  Local assessment: Week 12, Cycle 1 | 0.44 (0.56)
  Local assessment: Week 12, Cycle 2: number analyzed (Participants) | 125
  Local assessment: Week 12, Cycle 2 | 0.55 (0.65)
  Local assessment: Last study visit: number analyzed (Participants) | 147
  Local assessment: Last study visit | 0.53 (0.63)
  Central assessment: Week 12, Cycle 1: number analyzed (Participants) | 53
  Central assessment: Week 12, Cycle 1 | 0.08 (0.49)
  Central assessment: Week 12, Cycle 2: number analyzed (Participants) | 47
  Central assessment: Week 12, Cycle 2 | 0.18 (0.61)
  Central assessment: Last study visit: number analyzed (Participants) | 55
  Central assessment: Last study visit | 0.14 (0.59)

7. Secondary Outcome: Mean Change From Baseline in Maximal Walking Speed Barefoot at Week 12 of Each Treatment Cycle and at Last Study Visit
Description: The 10-meter walking speed test (WST) was used to measure active function in the LL. The participant performed the WST barefoot without a walking aid. If it was absolutely necessary that the participant used a cane, this may have been permitted provided that the same cane was used at baseline and all other walking speed assessments for that participant. The participant was given instructions to walk at his/her maximum speed. The time taken for the participant to walk from the start to the end of the 10 meters was recorded.
Time Frame: Week 12 of each treatment cycle and last study visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Dysport
Number analyzed (Participants) | 153
meters per second
  Week 12, Cycle 1: number analyzed (Participants) | 140
  Week 12, Cycle 1 | 0.081 (0.161)
  Week 12, Cycle 2: number analyzed (Participants) | 123
  Week 12, Cycle 2 | 0.116 (0.159)
  Last study visit: number analyzed (Participants) | 146
  Last study visit | 0.097 (0.187)

8. Secondary Outcome: Participant Satisfaction With the GSC at Week 6 and Week 12 of Each Treatment Cycle, Reinjection Cycle Visit and Last Study Visit
Description: Each participant received a personalised rehabilitation programme. The physiotherapist taught each participant the stretching postures and exercises to perform on a daily basis throughout the study. These were tailored to the individual participant's needs and formed the GSC therapy. The main focus was on the primary TT limb and then the other limb. Participant satisfaction was determined by asking the question "How satisfied are you TODAY regarding the GSC?" Responses were recorded using a 5-level Likert scale, as follows: completely satisfied (+2), rather satisfied (+1), neither satisfied nor dissatisfied (0), rather dissatisfied (-1), and completely dissatisfied (-2).
Time Frame: At baseline (for participants who had GSC previously only), Week 6 and Week 12 of each treatment cycle, reinjection cycle visit and last study visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 153
units on a scale
  Baseline for non-naïve participants to GSC only: number analyzed (Participants) | 39
  Baseline for non-naïve participants to GSC only | 1.8 (0.5)
  Week 6, Cycle 1: number analyzed (Participants) | 149
  Week 6, Cycle 1 | 1.3 (0.9)
  Week 12, Cycle 1: number analyzed (Participants) | 146
  Week 12, Cycle 1 | 1.4 (0.8)
  Reinjection cycle visit: number analyzed (Participants) | 140
  Reinjection cycle visit | 1.4 (0.7)
  Week 6, Cycle 2: number analyzed (Participants) | 136
  Week 6, Cycle 2 | 1.4 (0.7)
  Week 12, Cycle 2: number analyzed (Participants) | 130
  Week 12, Cycle 2 | 1.4 (0.8)
  Last study visit | 1.4 (0.8)

9. Secondary Outcome: Change From Baseline in Participant's Beliefs That the GSC Will Help to Improve Functional Capacity at Week 6 and Week 12 of Each Treatment Cycle, Reinjection Cycle Visit and Last Study Visit
Description: Participants were asked the following question: "Do you believe that GSC will help to improve your arm and leg function?" Responses were recorded on a 5-level Likert scale, as follows: very true of what I believe (+2), somewhat true of what I believe (+1), no opinion/don't know (0), somewhat untrue of what I believe (-1), and very untrue of what I believe (-2).
Time Frame: Week 6 and Week 12 of each treatment cycle, reinjection cycle visit and last study visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 153
units on a scale
  Week 6, Cycle 1: number analyzed (Participants) | 149
  Week 6, Cycle 1 | -0.2 (0.9)
  Week 12, Cycle 1: number analyzed (Participants) | 146
  Week 12, Cycle 1 | -0.1 (0.8)
  Reinjection cycle visit: number analyzed (Participants) | 140
  Reinjection cycle visit | -0.2 (0.8)
  Week 6, Cycle 2: number analyzed (Participants) | 136
  Week 6, Cycle 2 | -0.1 (0.7)
  Week 12, Cycle 2: number analyzed (Participants) | 130
  Week 12, Cycle 2 | -0.3 (0.8)
  Last study visit | -0.2 (0.8)

10. Secondary Outcome: Change From Baseline in Physiotherapist's Beliefs That the GSC Will Help to Improve Functional Capacity at Week 6 and Week 12 of Each Treatment Cycle, Reinjection Cycle Visit and Last Study Visit
Description: Physiotherapists were asked the following question: "Do you believe that GSC will help to improve your patient's arm and leg function?" Responses were recorded on a 5-level Likert scale, as follows: very true of what I believe (+2), somewhat true of what I believe (+1), no opinion/don't know (0), somewhat untrue of what I believe (-1), and very untrue of what I believe (-2).
Time Frame: Week 6 and Week 12 of each treatment cycle, reinjection cycle visit and last study visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 153
units on a scale
  Week 6, Cycle 1: number analyzed (Participants) | 113
  Week 6, Cycle 1 | -0.2 (0.6)
  Week 12, Cycle 1: number analyzed (Participants) | 110
  Week 12, Cycle 1 | -0.2 (0.6)
  Reinjection cycle visit: number analyzed (Participants) | 105
  Reinjection cycle visit | -0.1 (0.6)
  Week 6, Cycle 2: number analyzed (Participants) | 101
  Week 6, Cycle 2 | -0.2 (0.6)
  Week 12, Cycle 2: number analyzed (Participants) | 96
  Week 12, Cycle 2 | -0.2 (0.6)
  Last study visit: number analyzed (Participants) | 117
  Last study visit | -0.2 (0.7)

11. Secondary Outcome: Percentage of Days Over Study Period When GSC Therapy Was Performed
Description: The investigator counted the number of days when GSC therapy was not performed since the last visit. Using the total number of study days and the total number of days when GSC therapy was not performed, the number of days when GSC was performed was calculated.
Time Frame: From baseline to end of the study, up to 280 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of study days
Arm/Group | Dysport
Number analyzed (Participants) | 153
percentage of study days | 92.80 (9.85)

12. Secondary Outcome: Global Assessment of Benefits of the Study Therapy
Description: A global assessment of the benefits of the study therapy was made by the investigator and the participant (or the caregiver). The participant's caregiver performed the global assessment only in those cases when the participant was not capable to do this. Participants were asked the following question: "How would you rate the overall response to study therapy since baseline?" Responses on the global assessment were recorded on a 5-level Likert scale, as follows: much better (+2), a bit better (+1), the same (0), a bit worse (-1), and much worse (-2).
Time Frame: At reinjection cycle visit (Week 12, 16 or 20) and last study visit (Week 24 or 40)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 153
units on a scale
  Investigator: Reinjection cycle visit: number analyzed (Participants) | 138
  Investigator: Reinjection cycle visit | 1.4 (0.6)
  Investigator: Last study visit: number analyzed (Participants) | 147
  Investigator: Last study visit | 1.3 (0.7)
  Participant: Reinjection cycle visit: number analyzed (Participants) | 139
  Participant: Reinjection cycle visit | 1.4 (0.6)
  Participant: Last study visit: number analyzed (Participants) | 148
  Participant: Last study visit | 1.4 (0.7)

13. Secondary Outcome: Number of Participants Satisfied With a Longer Interval Between 2 Treatment Cycles
Description: Participants who were not reinjected at Week 12 of a given cycle, recorded their satisfaction with a longer interval between 2 injections collected at the corresponding reinjection visit or the last cycle visit (Week 16 or Week 20 for each cycle). To assess this, the participants were asked the following question: "Are you satisfied with a longer interval between 2 injections?". The possible answers were: Yes, No or No opinion.
Time Frame: At reinjection cycle visit (Week 16 or 20) and last study visit (Week 24 or 40)
Population: The ITT population included all participants who were injected at least once with the study treatment, who received at least 1 day of GSC therapy during the study and for whom a primary TT limb had been defined. Results are presented for participants who were not reinjected at Week 12 of the given cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dysport
Number analyzed (Participants) | 153
Participants
  Reinjection cycle visit: number analyzed (Participants) | 70
  Reinjection cycle visit: Yes | 52
  Reinjection cycle visit: No | 6
  Reinjection cycle visit: No opinion | 12
  Reinjection cycle visit: Missing | 0
  Last study visit: number analyzed (Participants) | 74
  Last study visit: Yes | 42
  Last study visit: No | 14
  Last study visit: No opinion | 12
  Last study visit: Missing | 6

14. Secondary Outcome: Change From Baseline in European Quality of Life 5 Dimensions (EQ-5D-5L) Scores at Last Study Visit
Description: Participants were asked to complete EQ-5D-5L questionnaire to assess their current health status. The EQ-5D-5L was a generic, preference-based measure of health-related quality of life (QoL). Questions were answered based on how the participant was feeling "Today". The EQ-5D-5L consists of 2 parts: EQ-5D descriptive system and EQ VAS. The EQ-5D descriptive system included questions for each of the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The VAS recorded participant's self-rated health on a vertical 20-centimeter VAS where the endpoints were labelled "The best health you can imagine" and "The worst health you can imagine". The EQ-5D-5L questionnaire scores range from 0-100, where 0= worst self-perceived health and 100= best self-perceived health. Positive change from baseline indicates an improvement in QoL.
Time Frame: At last study visit (Week 24 or 40)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 153
units on a scale
  Mobility: Last study visit: number analyzed (Participants) | 145
  Mobility: Last study visit | -0.3 (0.8)
  Self-care: Last study visit: number analyzed (Participants) | 145
  Self-care: Last study visit | -0.0 (0.8)
  Usual activities: Last study visit: number analyzed (Participants) | 145
  Usual activities: Last study visit | -0.3 (1.0)
  Pain/discomfort: Last study visit: number analyzed (Participants) | 145
  Pain/discomfort: Last study visit | -0.3 (0.9)
  Anxiety/depression: Last study visit: number analyzed (Participants) | 145
  Anxiety/depression: Last study visit | -0.1 (0.9)
  EQ VAS: Last study visit: number analyzed (Participants) | 145
  EQ VAS: Last study visit | 4.27 (18.71)

15. Secondary Outcome: Change From Baseline in Short Form 12 (SF-12) Scales at Last Study Visit
Description: The SF-12 was a short form questionnaire survey consisting of 12 questions, which were a subset of the SF-36 health survey. Most of the questions were answered based on how the participant had felt over the previous 4 weeks. The SF-12 covers 8 domains, including physical functioning, role-physical, body pain, general health, vitality, social functioning, role-emotional and mental health. The SF-12 questionnaire survey scale ranges from 0-100, where 0= lowest level of health and 100= highest level of health. Positive change from baseline indicates an improvement in QoL.
Time Frame: At last study visit (Week 24 or 40)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport
Number analyzed (Participants) | 153
units on a scale
  Physical score: Last study visit: number analyzed (Participants) | 145
  Physical score: Last study visit | 3.985 (7.358)
  Mental score: Last study visit: number analyzed (Participants) | 145
  Mental score: Last study visit | -0.008 (9.631)

ADVERSE EVENTS:
Time Frame: From first injection of study treatment up to end of the study or early withdrawal, approximately 40 weeks.
Description: The safety population included all participants who were injected at least once with the study treatment.
Arm/Group | Dysport
All-Cause Mortality (participants affected / at risk) | 1/157
Serious Adverse Events (participants affected / at risk) | 19/157
Other Adverse Events (participants affected / at risk) | 72/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport (N=157)
Epilepsy (Nervous system disorders) | 2 (2)
Brain stem stroke (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Myasthenic syndrome (Nervous system disorders) | 1 (1)
Vith nerve paralysis (Nervous system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Intervertebral discitis (Infections and infestations) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport (N=157)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 2 (2)
Fatigue (General disorders) | 5 (5)
Asthenia (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 3 (3)
Injection site haematoma (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 10 (12)
Contusion (Injury, poisoning and procedural complications) | 4 (9)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Diplopia (Eye disorders) | 2 (2)
Photopsia (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 2 (3)
Weight decreased (Investigations) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Injection site rash (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Therapeutic product ineffective (General disorders) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (2)
Clonic convulsion (Nervous system disorders) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Slow speech (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Angiogram abnormal (Investigations) | 1 (1)
ECG signs of myocardial ischaemia (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Abscess drainage (Surgical and medical procedures) | 1 (1)
Dental implantation (Surgical and medical procedures) | 1 (1)
Sinus operation (Surgical and medical procedures) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Thyroid disorder (Endocrine disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT02969356/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT02969356/SAP_001.pdf